CLINICAL TRIAL: NCT03751150
Title: Effectiveness of Injury Prevention Guidelines in Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Pia Desai, Doctoral Student, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SahgrenskaUH
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Sports Injury
Keywords: Running-related injury
MeSH Terms: conditions — Athletic Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Normal training, no intervention
- Intervention INT (Experimental): The intervention consists of an exercise program developed by a team specialised in orthopaedics, physiotherapy and biomechanics, based on the results from a recent prospective study in Gothenburg, Sweden. The exercises included cover muscle control training for the core, abductors, quadriceps and foot pronators, as well as foamrolling for the abductors, quadriceps, hamstrings, calf muscles and gluteal muscles. The runners will be instructed to perform the training program twice a week for the entire intervention period.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — The runners will be asked to perform the training program twice a week. The intervention consist of muscle control and foam rolling exercises for the lower extremities.
  Arms: Intervention INT

SUMMARY:
The aim of this trial is to investigate the effectiveness of specific training programs on the incidence of injuries in recreational runners. 408 runners between the ages of 18 and 55 years, will be recruited and randomly allocated to either the intervention group or control group. The intervention group will perform the training program twice a week in addition to their regular training. Injury data will be collected as the injuries occur and documentation of injury will follow a predetermined definition of injury. Participants will submit weekly reports of their running distance, frequency, running-related pain, as well as successful performance of the assigned training program for the intervention groups. The primary outcome is the incidence of injuries in all groups.

DETAILED DESCRIPTION:
Injuries and especially overuse injuries within recreational running are a common occurrence with higher incidence rates in novice runners but also in recreational runners training for a specific event. The mechanisms behind overuse injury development are thought to be multifactorial and certain parameters have shown to increase injury risk in recreational runners. The aim of this trial is to target these specific parameters and implement training programs to which recreational runners will adhere for a period of 18 weeks. About 408 male and female recreational runners, aged 18-55 years will be randomly allocated to one either the intervention (INT) or Control (CON).The INT group will perform an exercise program containing muscle control and foamrolling exercises in addition to their regular training, twice a week. The CON group will continue as per usual with their training. Training data will be collected on a weekly basis from all groups and pain and injury information will be submitted by the participants upon occurrence. The primary outcome measure is the number of sustained injuries in both groups. Participants will be recruited in December 2018 and the intervention will start in January 2019 for a period of 18 weeks, ending in May 2019. Data analyses are anticipated to be completed in September 2019.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female recreational runners with an average weekly running distance of at least 15km.

Exclusion Criteria:

* Injury to the lower extremities during the past 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Injury occurence | 18 weeks
  Incidence of running-related injuries

CONTACTS AND LOCATIONS:
Overall Officials: Jòn Karlsson, Prof, Study Chair — Sahlgrenska University Hospital; Stefan Grau, Prof, Study Director — Göteborg University
Locations (1):
- Cenrte for Health and Performance, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No